CLINICAL TRIAL: NCT05828602
Title: Feasibility of Pulmonary Rehabilitation Through Tele Rehabilitation Versus Traditional Center Based Pulmonary Rehabilitation for COPD in Pakistan
Brief Title: Pulmonary Rehabilitation Through Tele Rehabilitation for COPD in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rec/01373 Mehwish Haider
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator)
  Interventions: Other: Conventional treatment
- TeleRehabilitation (Experimental)
  Interventions: Other: TeleRehabilitation

INTERVENTIONS:
Other: Conventional treatment — Conventional treatment
  Arms: Conventional treatment
Other: TeleRehabilitation — TeleRehabilitation
  Arms: TeleRehabilitation

SUMMARY:
To determine the feasibility of Tele-rehabilitation vs traditional center-based pulmonary rehabilitation for people with chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* have a primary diagnosis of a chronic obstructive pulmonary disease
* aged ≥40 years
* be able to read and speak Urdu
* Vitally stable
* both gender

Exclusion Criteria:

* Inability to use technology, inadequate home setting, and patient's refusal.
* pulmonary hypertension or lung cancer attended pulmonary rehabilitation within the previous 18 months and had no hospitalizations for a respiratory cause since rehabilitation completion
* oxygen desaturation resulting in cessation of cardiopulmonary exercise testing (e.g. SpO2 < 80% during exercise on cycle ergometer)
* to ensure safety of unsupervised training
* unstable or brittle asthma with a hospital admission or emergency department presentation within the preceding 3 months, to ensure safety of unsupervised training
* co-morbidities which preclude exercise training, such as neurological or musculoskeletal impairment
* unable to follow verbal instructions, suffer from cognitive impairment, or have language difficulties

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Chronic respiratory questionnaire | 40 Days
  The chronic respiratory questionnaire has 20 items spread over four domains:
  dyspnea (5 items), tiredness (4 items), emotional function (7 items), and mastery. It can be administered by an interviewer or self-administered (4 items). Patients complete a 7-point rating scale on this form, with 1 being the worst possible experience and 7 being the best possible one (no impairment)
Physical activity via IPAQ | 40 Days
  Any voluntary skeletal muscle-driven movement that involves an energy cost is referred to as physical activity. All activities, regardless of intensity or time of day or night, can be considered physical activity. Both physical activity and unplanned activities incorporated into everyday routines are included . International Physical Activity Questionnaire short from will be utilized to measure level of physical activity. It consists of 7 items which ask about the activity of the last 7 days
Quality of life - Sf 12 | 40 Days
  The World Health Organization defines quality of life as "a person's view of their place in life in relation to their objectives, aspirations, standards, and concerns in the context of the culture and value systems in which they live." (20) . QOL will be assess via SF-12 Questionnaire. The SF-12 is a self-reported outcome measure that evaluates how one's health affects their day-to-day activities
Body mass index | 40 Days
  The body mass index (BMI) is a measurement that is based on a person's height and weight. The BMI is calculated by dividing the body weight by the square of the height, and it is expressed in kilograms per square meter (kg/m2) since weight is measured in kilograms and height is measured in meters
Borg Scale | 40 Days
  It is generally recognised that the Borg rating of perceived exertion scale is a reliable tool for determining perceived effort for a range of exercise modalities. The Borg scale (6-20) is intended to provide you with an approximation of your degree of effort based on your real heart rate when exercising. To determine your predicted heart rate, multiply your RPE by 10
Level of satisfaction scale | 40 Days
  It is a question that ranges from one extreme attitude to another using a 5 or 7- point scale that is sometimes referred to as a satisfaction scale. Very satisfied, Satisfied, Neither satisfied nor unsatisfied, Dissatisfied, and Very dissatisfied are examples of common responses on a 5-point Likert scale used to gauge satisfaction
Self-Structure open ended Questions | 40 Days
  Self-structured questionnaire was designed after reviewing the literature and with the help of experts in the field. it includes open ended questions, These questions will be asked in interview form from both the groups i.e Traditional Center Based Pulmonary Rehabilitation group and Tele Rehabilitation group, in which views on exercise, disease education, social contact, activity, accessibility, and support for participation will be assessed. This self-structured questionnaire will be a type of cognitive interview from both the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Hayatabad Medical Complex, Peshawar, Khyber PkahtoonKhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No